CLINICAL TRIAL: NCT02610322
Title: A Randomized Controlled Trial of Whole Soy Diet in Place of Red/Processed Meat and High Fat Dairy Products on Metabolic Features in Postmenopausal Women
Brief Title: Whole Soy Replacement Diet on Metabolic Features
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Liu Zhaomin, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRE-2013.121
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole soy group (Experimental): Whole soy replacement diet: to incorporate 4 servings of whole soy foods (equivalent to 25g soy protein) into their daily diet and reduce high saturated fat and cholesterol rich animal foods.
  Interventions: Behavioral: Whole soy replacement diet
- Control group (Placebo Comparator): Usual diet: to receive a conventional lifestyle education on MetS.
  Interventions: Behavioral: usual diet

INTERVENTIONS:
Behavioral: Whole soy replacement diet — Participants who are allocated to Whole soy group will receive a 30~40 min counseling session by an experienced nutritionist on: 1) conventional lifestyle education on metabolic syndrome (MetS); 2) The benefits of whole soy diet; 2) Practical techniques to incorporate of 4 servings of whole soy foods (equivalent to 25g soy protein) into their daily diet and reduce high saturated fat and cholesterol rich animal foods based on their prior 7-day dietary record during run-in; (3) Participants will also receive a pamphlet and an 30 min DVD which will provide practical cooking recipes with both illustration and demonstration on how to prepare whole soy foods/diet in an easy and fun way to replace fatty animal meat and dairy products
  Arms: Whole soy group
Behavioral: usual diet — Participants who are assigned to the usual diet group (control group) will receive a 5~10 min conventional lifestyle education on MetS by a research staff in which the general recommendation for macronutrient composition of the control diet will be 50-60% of energy as carbohydrate, 15-20% of energy as protein, and <30% of energy as total fat.
  Arms: Control group

SUMMARY:
Project title: A randomized controlled trial of whole soy diet in place of red/processed meat and high fat dairy products on metabolic features in postmenopausal women Objectives: Metabolic syndrome (MetS) is an escalating public health problem especially in postmenopausal women. Traditional whole soy foods are rich in unsaturated fats, high quality plant protein and various bioactive phytochemicals that could benefit on MetS. The aim of the study is to examine the effect of whole soy replacement diet on the features of MetS among postmenopausal women.

Hypothesis to be tested: Whole soy diet in place of red or processed meat and high fat dairy products will significantly improve metabolic features.

Design and subjects: This will be a 12-month randomized, single-blind, controlled trial among 208 postmenopausal women with high risk of MetS or early MetS.

Study instruments: After 4 weeks' run-in, participants will be randomly allocated to either of two intervention groups, whole soy replacement group or control group, each for 6 months.

Interventions: Subjects in whole soy group will be required to include 4 servings of whole soy foods (containing 25g soy protein) into their daily diet isocalorically replacing red or processed meat and high fat dairy products. Subjects in the control group will remain an usual diet.

Main outcome measures: The outcome measures will include the indices of metabolic features as well as a 10-year risk for ischemic cardiovascular disease.

Data analysis: The changes and %change of the metabolic features at 6- and 12-month will be compared among the two groups.

Expected results: Whole soy diet substitution of high saturated fat and cholesterol rich animal products will notably decrease the risk of MetS.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 45~70y within 15 years after menopause;
2. Participants who meet 2 or more of the following items:

   * waist circumference WC ≥80 cm;
   * triglyceride concentration ≥1.7 mmol/l;
   * HDL-c <50 mg/dl (1.29 mmol/l);
   * SBP/DBP ≥130/85 mm Hg;
   * fasting glucose ≥5.6 mmol/l.

Exclusion Criteria:

1. On use of medications known to affect body weight, lipids and glucose within past 3-month;
2. Medical history or presence of severe systemic or endocrine diseases;
3. Present or history of breast, endometrial or ovarian cancer;
4. Abnormal uterine bleeding after menopause;
5. On prescribed or vegetarian diet;
6. Known soy allergy.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of metabolic components of MetS (body weight, waist circumference, blood pressure, serum lipids and fasting glucose). | Will be measured at baseline, 6-month and 12-month after intervention.

SECONDARY OUTCOMES:
Changes of 10-year risk for ischemic cardiovascular disease (ICVD) | Will be assessed at baseline and 12-month after intervention.

REFERENCES:
- [Derived] Liu ZM, Ho S, Hao YT, Chen YM, Woo J, Wong SY, He Q, Xie YJ, Tse LA, Chen B, Su XF, Lao XQ, Wong C, Chan R, Ling WH. Randomised controlled trial of effect of whole soy replacement diet on features of metabolic syndrome in postmenopausal women: study protocol. BMJ Open. 2016 Sep 27;6(9):e012741. doi: 10.1136/bmjopen-2016-012741. PMID 27678545